CLINICAL TRIAL: NCT07309094
Title: Clinical, Morphometric and Biochemical Effects on Adiposopathy Associated With the Use of GLP-1 Receptor Agonists in Chronic Kidney Disease
Brief Title: Clinical, Morphometric and Biochemical Effects on Adiposopathy Associated With the Use of GLP-1RA in CKD
Acronym: ADIPO-CKD
Status: Recruiting | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Ana Checa-Ros, Co-PI. PhD Lecturer, Cardenal Herrera University
Other Study IDs: 23/424
Record Dates: First submitted 2025-12-03; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2; Obesity; Diabetes Mellitus, Type 2
Keywords: chronic kidney disease; type 2 diabetes mellitus; GLP-1RA; adiposopathy; perivisceral adipose tissue; perirenal adipose tissue; inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity; Diabetes Mellitus, Type 2; Inflammation | interventions — semaglutide; Liraglutide; dulaglutide; Exenatide; Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin; Canagliflozin; Tirzepatide; Angiotensin-Converting Enzyme Inhibitors; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples Serum samples Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- GLP-1RA Cohort: Patients receiving GLP-1RA, mainly semaglutide: weekly administration, subcutaneous form, from 0.25mg (starting dose) to 1mg (maintenance dose) with monthly increase (0.25-0.5-1mg)
  Interventions: Drug: GLP-1 receptor agonist; Drug: SGLT2 inhibitor
- SGLT2i Cohort: There will also be another comparative group of patients under SGLT2i
  Interventions: Drug: GLP-1 receptor agonist; Drug: SGLT2 inhibitor
- Other treatments: Patients not under SGLT2i or GLP-1RA/Tirzepatide influence, but receiving other treatments that are part of CKD and diabetes standard care
- Dual GIP GLP-1RA: Patients receiving tirzepatide: weekly administration, subcutaneous form, starting dose 2.5mg, maintenance 5mg
  Interventions: Drug: Tirzepatide; Drug: Other drugs

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Semaglutide: weekly subcutaneous administration, starting dose 0.25mg, maintenance dose 1mg
  Other Names: semaglutide; liraglutide; dulaglutide; exenatide
  Groups: GLP-1RA Cohort; SGLT2i Cohort
Drug: SGLT2 inhibitor — dapagliflozin: oral administration from 5 to 10mg/day
  Other Names: dapagliflozin; empagliflozin; canagliflozin
  Groups: GLP-1RA Cohort; SGLT2i Cohort
Drug: Tirzepatide — subcutaneous injection: starting dose 2.5 mg, maintenance 5mg (weekly administration)
  Groups: Dual GIP GLP-1RA
Drug: Other drugs — Patients not under SGLT2i or GLP-1RA influence, but receiving other treatments which are part of CKD standard care: mineralocorticoid receptor agonists, metformin, ACE inhibitors, ARBs...
  Other Names: ARBs; ACE inhibitors; Metformin; DPP4i; non steroidal mineralocorticoid receptor agonists
  Groups: Dual GIP GLP-1RA

SUMMARY:
Chronic kidney disease (CKD) is the progressive damage to kidney function, associated with an increased risk of cardiovascular diseases, such as stroke or myocardial infarct, particularly in the most severe stages of CKD, in which the patient requires dialysis. Several risk factors are reported for CKD, such as diabetes mellitus, obesity and hypertension. One of the most increasingly recognized risk factors is the fat tissue malfunction, known as adiposopathy. The accumulation of fat tissue around the organs in conditions of obesity or diabetes accelerates the production of pro-inflammatory factors that may worsen the kidney and heart damage. New antidiabetic medications, such as glucagon-like peptide-1 receptor agonists (GLP-1RA), have proven beneficial effects on the kidney and heart due to several mechanisms, including anti-inflammatory actions and a potential action on the fat tissue.

The aim of this study is to assess the link between adiposopathy and CKD, by investigating the changes in adiposopathy measures throughout treatment with GLP-1RA to a sample of patients with CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is defined as an irreversible abnormality of kidney structure and/or function lasting for more than three months. CKD is a major global health burden, affecting over 10% of the worldwide population and representing a leading cause of morbidity and mortality. Its progression to end-stage kidney disease (ESKD) drastically increases cardiovascular risk and is associated with a five-year survival rate of only approximately 50%. The principal risk factors for CKD-hypertension, obesity and type 2 diabetes (T2DM) in particular-are intrinsically linked through the dysfunction of fat/adipose tissue (AT), also known as adiposopathy.

Adiposopathy is a key driver of cardiorenal risk in CKD. Evidence from bioimpedance, imaging techniques (CT, MRI), and molecular biology studies confirm that alterations in adipose tissue-including its quantity, distribution (e.g., perirenal, epicardial), radiodensity, and the secretion of pro-inflammatory adipokines-are powerful triggers of cardiorenal damage and mortality in these patients. This understanding frames obesity, T2DM, cardiovascular diseases (CVDs), and CKD as different manifestations of a shared spectrum, now termed adiposity-based chronic disease (ABCD), necessitating an "adipocentric" therapeutic approach.

One hallmark feature of adiposopathy is the reprogramming and increase in size of certain region-specific adipose tissue. Perivisceral adipose tissue plays a pivotal role in adiposity-based chronic diseases as it releases adipokines and cytokines that not only contribute to the systemic pro-inflammatory and oxidative stress processes but may also influence the function of the organs surrounded by this tissue.

GLP-1RA stimulates the receptor for glucagon-like peptide-1 (GLP-1), an incretin-like hormone released in the large intestine that reduces serum glucose concentrations by stimulating the glucose-dependent release of insulin, inhibiting the hypersecretion of glucagon (except in hypoglycemia periods) and promoting satiety. GLP-1RA reduced the incidence of cardiovascular death in patients with T2DM compared with placebo and decreased the incidence of major kidney events, also reducing the progression of kidney dysfunction and the risk of death. In animals, the observed morphological changes generated by GLP-1RA could be underlined by potential actions on adipose tissue remodeling, as these drugs upregulated the expression of AT-browning related genes in perivisceral white adipose tissue from murine models, although the transcriptomic effects from GLP-1RA on the adiposopathy process are still unknown.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age
* diagnosed with CKD in stages G1, G2, G3a, G3b, and G4, not candidate for dialysis
* had uncontrolled T2DM, CVDs and/or obesity
* willing to participate in the study and sign informed consent

Exclusion Criteria:

* Age <18 years
* pregnancy
* CKD in stage G5 or G4 candidate for dialysis
* neuropsychiatric diseases preventing the patient from understanding the benefits/risks associated with the project
* refusal to participate and/or consent revocation were considered as exclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be assigned to the different groups according to current treatment criteria:
  SGLT2i: patients with CKD and T2DM with an eGFR ≥20ml/min/1.73m2; patients with CKD and eGFR ≥20ml/min/1.73m2, accompanied by an urinary albumin-to-creatinine ratio (ACR) ≥200mg/g; patients with CKD and heart failure, irrespective of level of albuminuria; or subjects with CKD and eGFR 20-45ml/min/1.73m2, with ACR <200mg/g.
  GLP-1RA/tirzepatide: In patients with T2D and CKD who have not achieved individualized glycemic targets despite use of metformin and SGLT2i treatment, or who are unable to use those medications.
  Other treatments: patients not meeting the criteria to be treated with SGLT2i or GLP-1RA/tirzepatide
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography change in perirenal adipose tissue thickness | 16 months
  Change in perirenal adipose tissue thickness as measured with ultrasonography
Change in estimated glomerular filtration rate | 16 months
  Change in eGFR as per the CKD-EPI formula

SECONDARY OUTCOMES:
Ultrasonographic Change in epicardial adipose tissue thickness | 16 months
  Change in epicardial adipose tissue thickness as measured with ultrasonography
Change in serum leptin levels | 16 months
  Serum leptin levels measured with proteomic analysis
Change in visceral fat area | 16 months
  Changes in visceral fat area (cm2) as measured with body composition measures (bioimpedance)
Ultrasonographic Change in subcutaneous adipose tissue | 16 months
  Change in subcutaneous adipose tissue thickness as measured with ultrasonography
Ultrasonographic Change in preperitoneal adipose tissue thickness | 16 months
  Change in preperitoneal adipose tissue thickness as measured with ultrasonography
Ultrasonographic Change in intrahepatic adipose tissue | 16 months
  Change in intrahepatic adipose tissue echogenicity
Change in subcutaneous fat area | 16 months
  Change in subcutaneous fat area (cm2) as measured with bioimpedance
Changes in muscle mass (kg) | 16 months
  Changes in muscle mass as measured with bioimpedance
Change in serum adiponectin levels | 16 months
  Serum adiponectin levels measured with proteomic analysis
Change in urinary levels of Kidney Injury Molecule-1 | 16 months
  Change in urinary levels of KIM-1 measured with ELISA, as an early marker of kidney damage

OTHER OUTCOMES:
Change in systemic inflammation markers | 16 months
  Change in serum C-reactive protein levels
Change in systemic inflammation markers | 16 months
  Change in serum interleukin-6 levels
Change in systemic inflammation markers | 16 months
  Change in serum tumor necrosis factor-alpha levels

CONTACTS AND LOCATIONS:
Overall Officials: Luis D'Marco, MD, PhD, Principal Investigator — Cardenal Herrera University; Ana Checa-Ros, MD, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Vithas Valencia Consuelo, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Due to ethical restrictions and in accordance with General Protection Data Regulation, no identifiable patient information will be shared.

REFERENCES:
- [Background] Zhao L, Li W, Zhang P, Wang D, Yang L, Yuan G. Liraglutide induced browning of visceral white adipose through regulation of miRNAs in high-fat-diet-induced obese mice. Endocrine. 2024 Jul;85(1):222-232. doi: 10.1007/s12020-024-03734-2. Epub 2024 Feb 20. PMID 38378894
- [Background] Ying Y, Zhu H, Liang Z, Ma X, Li S. GLP1 protects cardiomyocytes from palmitate-induced apoptosis via Akt/GSK3b/b-catenin pathway. J Mol Endocrinol. 2015 Dec;55(3):245-62. doi: 10.1530/JME-15-0155. Epub 2015 Sep 18. PMID 26386043
- [Background] Carraro-Lacroix LR, Malnic G, Girardi AC. Regulation of Na+/H+ exchanger NHE3 by glucagon-like peptide 1 receptor agonist exendin-4 in renal proximal tubule cells. Am J Physiol Renal Physiol. 2009 Dec;297(6):F1647-55. doi: 10.1152/ajprenal.00082.2009. Epub 2009 Sep 23. PMID 19776173
- [Background] Perkovic V, Tuttle KR, Rossing P, Mahaffey KW, Mann JFE, Bakris G, Baeres FMM, Idorn T, Bosch-Traberg H, Lausvig NL, Pratley R; FLOW Trial Committees and Investigators. Effects of Semaglutide on Chronic Kidney Disease in Patients with Type 2 Diabetes. N Engl J Med. 2024 Jul 11;391(2):109-121. doi: 10.1056/NEJMoa2403347. Epub 2024 May 24. PMID 38785209
- [Background] Giugliano D, Maiorino MI, Bellastella G, Longo M, Chiodini P, Esposito K. GLP-1 receptor agonists for prevention of cardiorenal outcomes in type 2 diabetes: An updated meta-analysis including the REWIND and PIONEER 6 trials. Diabetes Obes Metab. 2019 Nov;21(11):2576-2580. doi: 10.1111/dom.13847. Epub 2019 Aug 28. PMID 31373167
- [Background] D'Marco L, Puchades MJ, Panizo N, Romero-Parra M, Gandia L, Gimenez-Civera E, Perez-Bernat E, Gonzalez-Rico M, Gorriz JL. Cardiorenal Fat: A Cardiovascular Risk Factor With Implications in Chronic Kidney Disease. Front Med (Lausanne). 2021 May 25;8:640814. doi: 10.3389/fmed.2021.640814. eCollection 2021. PMID 34113631
- [Background] Ku E, Lee BJ, Wei J, Weir MR. Hypertension in CKD: Core Curriculum 2019. Am J Kidney Dis. 2019 Jul;74(1):120-131. doi: 10.1053/j.ajkd.2018.12.044. Epub 2019 Mar 19. PMID 30898362
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Khan MZ, Syed M, Osman M, Faisaluddin M, Sulaiman S, Farjo PD, Khan MU, Agrawal P, Alharbi A, Khan SU, Munir MB, Balla S. Contemporary Trends and Outcomes in Patients With ST-Segment Elevation Myocardial Infarction and End-Stage Renal Disease on Dialysis: Insight from the National Inpatient Sample. Cardiovasc Revasc Med. 2020 Dec;21(12):1474-1481. doi: 10.1016/j.carrev.2020.05.004. Epub 2020 May 11. PMID 32444271
- [Background] Moisi MI, Bungau SG, Vesa CM, Diaconu CC, Behl T, Stoicescu M, Toma MM, Bustea C, Sava C, Popescu MI. Framing Cause-Effect Relationship of Acute Coronary Syndrome in Patients with Chronic Kidney Disease. Diagnostics (Basel). 2021 Aug 23;11(8):1518. doi: 10.3390/diagnostics11081518. PMID 34441451
- [Background] Artzi-Medvedik R, Kob R, Fabbietti P, Lattanzio F, Corsonello A, Melzer Y, Roller-Wirnsberger R, Wirnsberger G, Mattace-Raso F, Tap L, Gil P, Martinez SL, Formiga F, Moreno-Gonzalez R, Kostka T, Guligowska A, Arnlov J, Carlsson AC, Freiberger E, Melzer I; SCOPE investigators. Impaired kidney function is associated with lower quality of life among community-dwelling older adults : The screening for CKD among older people across Europe (SCOPE) study. BMC Geriatr. 2020 Oct 2;20(Suppl 1):340. doi: 10.1186/s12877-020-01697-3. PMID 33008306
- [Background] George LK, Koshy SKG, Molnar MZ, Thomas F, Lu JL, Kalantar-Zadeh K, Kovesdy CP. Heart Failure Increases the Risk of Adverse Renal Outcomes in Patients With Normal Kidney Function. Circ Heart Fail. 2017 Aug;10(8):e003825. doi: 10.1161/CIRCHEARTFAILURE.116.003825. PMID 28765150
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Foreman KJ, Marquez N, Dolgert A, Fukutaki K, Fullman N, McGaughey M, Pletcher MA, Smith AE, Tang K, Yuan CW, Brown JC, Friedman J, He J, Heuton KR, Holmberg M, Patel DJ, Reidy P, Carter A, Cercy K, Chapin A, Douwes-Schultz D, Frank T, Goettsch F, Liu PY, Nandakumar V, Reitsma MB, Reuter V, Sadat N, Sorensen RJD, Srinivasan V, Updike RL, York H, Lopez AD, Lozano R, Lim SS, Mokdad AH, Vollset SE, Murray CJL. Forecasting life expectancy, years of life lost, and all-cause and cause-specific mortality for 250 causes of death: reference and alternative scenarios for 2016-40 for 195 countries and territories. Lancet. 2018 Nov 10;392(10159):2052-2090. doi: 10.1016/S0140-6736(18)31694-5. Epub 2018 Oct 16. PMID 30340847
- [Background] Borg R, Carlson N, Sondergaard J, Persson F. The Growing Challenge of Chronic Kidney Disease: An Overview of Current Knowledge. Int J Nephrol. 2023 Mar 1;2023:9609266. doi: 10.1155/2023/9609266. eCollection 2023. PMID 36908289
- See also: Research group website — http://www.uchceu.es/grupos-lineas-investigacion/investigacion-de-enfermedades-cardiorenales-y-metabolicas-idecam
- Available data/document: Statistical Analysis Plan — http://osf.io/
- Available data/document: Analytic Code — http://osf.io